CLINICAL TRIAL: NCT05204056
Title: Application of Iced Normal Saline Combined With Cocktail Perfusion in Total Knee Arthroplasty: Randomized Controlled Trial
Brief Title: Application of Iced Normal Saline Combined With Cocktail Perfusion in Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yantai Yuhuangding Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2018-149
Record Dates: First submitted 2022-01-10; First posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Pain, Postoperative; Blood Loss, Postoperative
MeSH Terms: conditions — Pain, Postoperative; Postoperative Hemorrhage | interventions — Tranexamic Acid; Morphine; Epinephrine; Perfusion

STUDY DESIGN:
Intervention Model Description: Recruited patients were divided into three groups with different recipes. Group A: twenty patients who were given intraoperative joint cavity infusion therapy using 20ml tranexamic and 40ml iced normal saline; Group B twenty patients who were given 20ml of iced normal saline, 20ml of iced cocktail and 20ml of tranexamic; the left twenty patients were given joint cavity infusion therapy with 20ml tranexamic only as the control group. Intravertebral anaesthesia was selected for the surgery and the operations were performed by the same surgical team. The average operation time was about 1.5 hours, which lasted from the compression of the tourniquet to completed wound dressing.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Twenty patients who were given intraoperative joint cavity infusion therapy using 20ml tranexamic and 40ml iced normal saline.
  Interventions: Drug: iced normal saline; Drug: Tranexamic acid injection
- Group B (Experimental): Twenty patients who were given 20ml of iced normal saline, 20ml of iced cocktail and 20ml of tranexamic
  Interventions: Drug: iced normal saline; Drug: Tranexamic acid injection; Other: Cocktail (composing by Ropivacaine, Morphine and Epinephrine) perfusion
- Control group (Active Comparator): Twenty patients were given joint cavity infusion therapy with 20ml tranexamic only as the control group
  Interventions: Drug: Tranexamic acid injection

INTERVENTIONS:
Drug: iced normal saline — Iced normal saline (20ml) was given intraoperative joint cavity infusion therapy
  Other Names: H19983149
  Arms: Group A; Group B
Drug: Tranexamic acid injection — 20ml of tranexamic was given with iced normal saline for intraoperative joint cavity infusion.
  Other Names: H43020565
Other: Cocktail (composing by Ropivacaine, Morphine and Epinephrine) perfusion — Cocktail was formulated during the operation by mixing Ropivacaine 150mg, Morphine 10mg and Epinephrine 1mg, then normal saline was used to dilute the mixture to 60ml. Then the cocktail mixture was applied for the joint cavity perfusion.
  Arms: Group B

SUMMARY:
Sixty patients undergoing TKA were divided into three groups, then three different intro-operative articular cavity perfusion treatment was given according to the randomized, double-blind and controlled rule. One way ANOVA analysis on visual analogue scale (VAS) score, functional recovery, drainage, and edema of the affected limb were performed to assess the efficiency of the treatment in the following three days after the operation.

DETAILED DESCRIPTION:
Patients with confirmed primary knee osteoarthritis in stage IV by preoperative X-ray were included in present study, whilst subsequent arthritis (including rheumatoid arthritis, Gouty arthritis, traumatic arthritis, etc.) were excluded. After assessment, sixty qualified patients who voluntarily participating in this study have understood the research project were included in the present study and the corresponding consent forms were signed. Patients were randomly classified into three groups with different interventions, each group contains 20 patients. Group A: twenty patients who were given intraoperative joint cavity infusion therapy using 20ml tranexamic and 40ml iced normal saline; Group B twenty patients who were given 20ml of iced normal saline, 20ml of iced cocktail and 20ml of tranexamic; the left twenty patients were given joint cavity infusion therapy with 20ml tranexamic only as the control group. All the study personnel including the patients, their family members, the nursing staff and the leading operator were blind to the treatment allocation.

ELIGIBILITY:
Inclusion Criteria:

Patients with confirmed primary knee osteoarthritis in stage IV by preoperative X-ray were included in present study. Kellgren-Lawrence Radiology standards for stage IV were listed as follows: obviously narrowed joint space; vast osteophytes are formed; severe osteosclerosis under the cartilage; bone hypertrophy and evident deformity

Exclusion Criteria:

Subsequent arthritis (including rheumatoid arthritis, Gouty arthritis, traumatic arthritis, etc.) were excluded.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Reduced pain | three days after operation
  the pain after operation reduced significantly.

SECONDARY OUTCOMES:
Reduced bleeding | 24 hours drainage.
  The blood loss reduced significantly after operation.

OTHER OUTCOMES:
increased HSS scores | 3 days after operation
  The HSS scores increased markedly after operation.

CONTACTS AND LOCATIONS:
Overall Officials: Laijian Sui, Doctor, Study Chair — Yantai Yuhuangding Hospital
Locations (1):
- Yantai Yuhuangding Hospital, Yantai, Shandong, China

IPD SHARING:
Plan to Share IPD: No